CLINICAL TRIAL: NCT01847027
Title: Phase 2 Study of the Effect of a Nutritional Supplement and Exercise on Human Stem Cells
Brief Title: Exercise and NutraStem (NT-020): Effects on Stem Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, Meharvan Singh, Professor, Department of Pharmacology and Neuroscience, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-162
Record Dates: First submitted 2013-05-01; First posted 2013-05-06 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Adult Stem Cell Proliferation
Keywords: Healthy; Stem cells; Aging; Increase stem cell replacement; decreased stem cell proliferation
MeSH Terms: interventions — NT020 formula; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active supplement (Active Comparator): NutraStem, 2 tablets daily, Vitamin D3 (2000 IU), BioVin® (40 mg) and the proprietary blend (900mg).
  Interventions: Drug: NutraStem
- Sugar pill (Placebo Comparator): The placebo is identical in appearance to the NutraStem® supplement and contains the following ingredients in a Vegi Capsule:
  MCC200 DICALCIUM PHOSPHATE BROWN LAKE BLEND (SENSIENT # 09127 ) RED DYE DB-088 (COLORCON) MAGNESIUM STEARATE BLUE #1 ALUM LAKE (POWDER)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NutraStem — Determine whether NutraStem® in combination with an exercise stimulus will cause increased human peripheral blood sample levels of CD34+ and CD133+ adult stem cells and whether these stem cells display more protection against oxidative stress.
  Determine whether NutraStem® in combination with an exercise stimulus will cause increased human peripheral blood sample levels of CD34+ and CD133+ adult stem cells and whether these stem cells display more protection against oxidative stress.
  Other Names: NT-020
  Arms: Active supplement
Drug: Placebo — Determine whether NutraStem® in combination with an exercise stimulus will cause increased human peripheral blood sample levels of CD34+ and CD133+ adult stem cells and whether these stem cells display more protection against oxidative stress.
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to see if an investigational supplement called NutraStem® will increase the amount of stem cells in human blood at rest and after exercise. The ingredients found in NutraStem® can be found in nutrition or vitamin shops/stores.

DETAILED DESCRIPTION:
A randomized double blinded placebo controlled trial of a nutraceutical preparation. Up to 60 men and women between the ages of 50 and 70, and generally healthy will participate in this study. . Up to 30 participants will receive the nutritional supplement and up to 30 will receive placebo.

Potential participants will be screened by telephone and have the study explained to them in detail. If they qualify and choose to participate they will come in for the first of three visits. Informed consent will be obtained and demographic information collected. Information requested on the demographic form includes ethnicity, income, education, marital status, smoking and alcohol use, and exercise habits. Next they will have blood pressure checked and if not within parameters they will be dropped from the study and informed that they need to follow up the abnormal result with their health care provider. Those that pass these screening tests will have 15 to 25 cc's of peripheral blood (serum) collected by the study coordinator via venipuncture while at rest. They will then stretch for 2 minutes (60 seconds marching in place followed by 10 toe touches) followed by accelerating treadmill walking exercise. The exercise intervention will consist of a 15 minute period of walking on a treadmill. The treadmill will not be inclined during the intervention. The participants target heart rate will be determined by deducting their age from 220. They will start walking on the treadmill at a speed of 1.7 mph and the speed will be titrated as indicated to keep their heart rate at 50 to 90% of target. Heart rate will be monitored via the pulse oximetry feature of the Welch Allyn vital signs monitor. Blood pressure will be measured every 3 minutes during the exercise intervention and until they have returned to baseline (within 10 points) following cessation of the exercise protocol. The test will be stopped for any participant complaint of chest pain, excess fatigue, difficulty breathing, a blood pressure reading of more than 180/94, or a participant request. If symptoms increase or do not completely resolve with 15 minutes of rest the study coordinator will call 911 (through campus police) to activate the EMS response. If symptoms resolve completely within 15 minutes participants will be withdrawn from the study and advised to follow up with their health care provider. Any participant unable to complete the exercise intervention for any reason will be withdrawn from the study.

Five to fifteen minutes after the exercise intervention has been completed blood will again be collected in exactly the same manner as the resting sample. Participants will then receive a 2 week supply of either NutraStem or placebo and will be advised to take one tablet every morning and evening before meals for the next 2 weeks. If the participant is unable to complete any portion of the visit activities at any visit they will be withdrawn from the study due to their inability to complete the study. All visit activities will be recorded in detail on the visit session record.

The second visit will occur 2 weeks later and include a blood pressure check, an at rest blood draw, the exercise intervention, and then a repeat blood draw five to fifteen minutes after completion of the intervention. Participants will then receive a 2 week supply of either NutraStem or placebo and will be advised to take one tablet every morning and evening before meals for the next 2 weeks. I Participants will be advised to bring their empty pill containers to their next session so we can confirm they are taking the supplement as required. If the blood pressure is outside of the specified range they will be dropped from the study and no blood collection or study intervention will take place.

The third visit will be the same as the second visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 50 to 70 years old
* Ability to walk on a treadmill for 15 minutes.

Exclusion Criteria:

* Age less than 50 or greater than 70 years of age.
* A history of difficult veins/difficulty obtaining blood samples
* Unwilling to follow the procedures of the trial
* Participated in more than 2 sessions per week of strenuous exercise in the last month
* Unable to tolerate the ingredients in NutraStem® or placebo, or have food allergies
* Intentionally lost or gained 10 or more pounds of body weight in the last 3 months
* Acute illness
* Severe co-morbid disease
* Use of any prescription or non-prescription products for antioxidant regimen or stem cell supplement within the past 4 weeks
* Diabetic
* Uncontrolled hypertension
* Recent cardiovascular event (past 36 months), or a family history of sudden death or heart attacks before the age of 55
* Body Mass Index (BMI) of less than 20 or greater than 35 m/kg2;
* Participated in a clinical trial in the past 4 weeks
* Take methadone, insulin, anticoagulants (blood thinners), MAO's or similar medications
* Anticipate the need for surgery of any type during the entire study;
* Plan to donate blood or blood products during the study or for thirty (30) days following the study
* Active peptic ulcer disease or reliable history of gastrointestinal bleeding within the past five (5) years
* Recurrent or a history of intestinal disorders that may interfere with the absorption of the product
* Any disease or condition that in the investigator's opinion compromises the integrity of the clinical trial or the safety of the subject

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meharvan Singh, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center - Center for Biohealth, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Supplement: NutraStem, 2 tablets daily, Vitamin D3 (2000 IU), BioVin® (40 mg) and the proprietary blend (900mg).
  NutraStem: Determine whether NutraStem® in combination with an exercise stimulus will cause increased human peripheral blood sample levels of CD34+ and CD133+ adult stem cells and whether these stem cells display more protection against oxidative stress.
  Determine whether NutraStem® in combination with an exercise stimulus will cause increased human peripheral blood sample levels of CD34+ and CD133+ adult stem cells and whether these stem cells display more protection against oxidative stress.
- Sugar Pill: The placebo is identical in appearance to the NutraStem® supplement and contains the following ingredients in a Vegi Capsule:
  MCC200 DICALCIUM PHOSPHATE BROWN LAKE BLEND (SENSIENT # 09127 ) RED DYE DB-088 (COLORCON) MAGNESIUM STEARATE BLUE #1 ALUM LAKE (POWDER)
  Placebo: Determine whether NutraStem® in combination with an exercise stimulus will cause increased human peripheral blood sample levels of CD34+ and CD133+ adult stem cells and whether these stem cells display more protection against oxidative stress.
Period: Overall Study
Arm/Group | Active Supplement | Sugar Pill
Started | 11 | 12
Completed | 10 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Supplement | Sugar Pill | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (6.3) | 59.5 (6.1) | 59.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of CD133+ Cells
Description: The percentage of CD133+ cells detected in blood samples
Time Frame: Baseline, 2 weeks, 4 weeks
Population: subjects who completed all three visits and from whom blood draws were obtained
Measure: Mean (Standard Deviation); unit: percent of total
Arm/Group | Active Supplement | Sugar Pill
Number analyzed (Participants) | 10 | 10
percent of total
  Baseline (visit 1) | 0.50 (0.39) | 0.28 (0.15)
  2 weeks (visit 2) | 0.54 (0.49) | 0.47 (0.54)
  4 weeks (visit 3) | 0.37 (0.25) | 0.35 (0.27)

2. Primary Outcome: Percent of CD34+ Cells
Description: Percent of CD34+ cells detected in blood samples
Time Frame: Baseline, 2 weeks, 4 weeks
Population: Subjects who completed all three visit and from whom blood draws were successful
Measure: Mean (Standard Deviation); unit: percent of total
Arm/Group | Active Supplement | Sugar Pill
Number analyzed (Participants) | 10 | 10
percent of total
  Baseline (visit 1) | 9.46 (6.98) | 14.31 (7.4)
  2 weeks (visit 2) | 7.64 (8.29) | 7.13 (3.97)
  4 weeks (visit 3) | 7.29 (6.08) | 8.49 (5.95)

3. Secondary Outcome: Markers of Oxidative Stress
Description: Blood levels of C reactive protein
Time Frame: Baseline, 4 weeks
Population: Subjects who completed all three visits
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Active Supplement | Sugar Pill
Number analyzed (Participants) | 10 | 10
ng/L
  Baseline (visit 1) | 1695848.62 (2084023.54) | 1843643.43 (1391654.22)
  4 weeks (visit 3) | 873777.84 (647730.33) | 1935423.36 (1096810.43)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Blood pressure is monitored in individuals while exercising (treadmill walking).
Arm/Group | Active Supplement | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Supplement (N=11) | Sugar Pill (N=12)
vasovagal response (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-01-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT01847027/Prot_SAP_ICF_000.pdf